CLINICAL TRIAL: NCT03410888
Title: Popliteal Approach to Sciatic Nerve Block Provides Postoperative Analgesia That Is Not Inferior to That of the Infragluteal Approach in Patients Undergoing Unilateral Total Knee Arthroplasty Under Spinal Anesthesia
Brief Title: Popliteal Approach to Sciatic Nerve Block Is Not Inferior to Infragluteal Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0306-B
Record Dates: First submitted 2013-02-11; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Neuromuscular Blockade
Keywords: sciatic nerve block; infragluteal approach; popliteal approach

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- popliteal approach (Experimental): Blockade of the sciatic nerve at the level of the popliteal fossa.
  Interventions: Procedure: Popliteal approach
- infragluteal approach (Active Comparator): Blocking the sciatic nerve at the subgluteal level.
  Interventions: Procedure: Infragluteal approach

INTERVENTIONS:
Procedure: Popliteal approach — Popliteal approach:
  Under ultrasound guidance a 50 to 90 mm 22 G needle is inserted in and advanced to contact the target nerve until nerve movement is detected. The end point of nerve block in this group is obtaining a circumferential local anesthetic spread around the sciatic nerve.
  Arms: popliteal approach
Procedure: Infragluteal approach — Infragluteal approach: The patients in this group will receive sciatic bock according to the approach described by Chan et al. Ultrasound scanning will be used to identify and mark the greater trochanter laterally and the ischial tuberosity medially. The sciatic nerve is usually found anterior (deep) to the gluteus maximus muscle and lateral to the origin of the biceps femoris muscle at the ischial tuberosity as well as medial to the greater trochanter. The end point of nerve block in this group is obtaining a circumferential local anesthetic spread around the sciatic nerve.
  Arms: infragluteal approach

SUMMARY:
Study Hypothesis The investigators approach to demonstrate noninferiority of analgesia provided by popliteal block in TKA surgery will be based on a hypothesis of absence of a clinically significant difference in pain visual analogue sores (VAS) between the analgesia provided by the popliteal block and that of the infragluteal sciatic block in TKA surgery patients.

DETAILED DESCRIPTION:
Sciatic nerve block provides clinically significant analgesic benefits following total knee arthroplasty (TKA). These benefits include a reduction in pain scores and decrease analgesic requirements.

Despite these benefits, sciatic nerve block has remained among the least performed peripheral nerve block by anesthesiologists. Some impediments relating to single shot sciatic nerve block (SSNB) that may cause anesthesiologists to avoid it include, patient discomfort due to needle passage through dense gluteal or thigh adipose and musculature, and unreliable success because of difficulty in localizing the sciatic nerve (particularly in obese patients).

Even in the current era of US guidance, sciatic nerve block remains a challenge. Despite its helpfulness, ultrasound technology remains hindered by an intrinsic limitation: a trade off between depth of penetration and image resolution; therefore, it works well for superficial blocks but becomes less useful when deep structures are imaged-ironically where this guidance is needed most. The challenge of anatomical depth, as in the case of the sciatic nerve, is one remaining challenge that dictates practical restrictions on the patterns of practice of ultrasound-guided regional anesthesia.

Actually, the recommendations of the Joint Committee for Education and Training composed of the American Society of Regional Anesthesia and the European Society of Regional Anesthesia cite the depth of block resulting in degradation of both ultrasound and needle image as the first among other causes that increase the level of difficulty of a nerve block.

As the sciatic nerve travels caudally in the body, it becomes more superficial with less thickness of tissue separating it from skin surface, making distal sciatic nerve block an attractive alternative. Indeed, both articular branches which provide sensory innervation to the knee joint as well as its muscular branches which provide innervation to the muscles surrounding knee joint most commonly arise from the sciatic nerve either at the knee level, or just above the knee or within the popliteal fossa.

Blockade of the sciatic nerve at the level of the popliteal fossa, commonly termed a popliteal block, is technically easier to perform than gluteal sciatic block and may even be associated with less risk of intravascular injection and nerve injury. Indeed, popliteal block has been reported to provide good postoperative analgesia in total knee replacement and other major knee surgery. However, the small posterior cutaneous nerve of the thigh, which supplies only the skin on the back of the thigh and knee, separates from the sciatic nerve proximally and variably in the gluteal region, and will be spared in more distal approaches. It is for this reason why many practitioners are hesitant to perform distal sciatic nerve blocks for TKA. However, the relative importance of the posterior cutaneous nerve of the thigh for post-operative analgesia following TKA is unknown and maybe clinically insignificant.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* American Society of Anesthesiologists (ASA) Physical Status Scale I-III patients undergoing unilateral TKA under spinal anesthesia and nerve blocks
* Ages 18-85
* BMI ≤ 38 kg/m2

Exclusion Criteria:

* Chronic pain disorders
* Significant pre-existing neurological deficits or peripheral neuropathy affecting the lower extremity
* Abuse of drugs or alcohol
* Allergies to any medication included in the study protocol
* Contraindication to spinal anesthesia or failure to institute spinal anesthesia after performing femoral and sciatic blocks
* Bilateral TKA surgeries
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain scores. The score at 6 hours will be considered as primary outcome. | 6 hours
  Overall pain level as well as pain localized o the back of the knee will be assessed at rest and on movement (knee flexion) and will be quantified with a 100 mm VAS pain scale score, with 0 representing no pain and 100 representing the worst imaginable pain.

SECONDARY OUTCOMES:
Sensory/Motor block onset assesment in the sciatic nerve distribution | 60 minutes
  The onset of sensory block will be assessed in the sciatic nerve distribution within 60 minutes of local anesthetic injection.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Allen HW, Liu SS, Ware PD, Nairn CS, Owens BD. Peripheral nerve blocks improve analgesia after total knee replacement surgery. Anesth Analg. 1998 Jul;87(1):93-7. doi: 10.1097/00000539-199807000-00020. PMID 9661553
- [Background] Cook P, Stevens J, Gaudron C. Comparing the effects of femoral nerve block versus femoral and sciatic nerve block on pain and opiate consumption after total knee arthroplasty. J Arthroplasty. 2003 Aug;18(5):583-6. doi: 10.1016/s0883-5403(03)00198-0. PMID 12934209
- [Background] Bailey SL, Parkinson SK, Little WL, Simmerman SR. Sciatic nerve block. A comparison of single versus double injection technique. Reg Anesth. 1994 Jan-Feb;19(1):9-13. PMID 8148303